CLINICAL TRIAL: NCT03681977
Title: The Influence of Medial Pivot Knee Arthroplasty Implant Design on Joint Mechanics, Muscle Activation and Clinical Outcomes
Brief Title: Clinical Outcomes of MP Persona vs. Persona Knee-PS
Acronym: MP-Persona
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Jewish General Hospital (Other); McGill University (Other); Zimmer Biomet (Industry); Montreal General Hospital (Other)
Responsible Party: Principal Investigator, John Antoniou, MD PhD, Principal Investigator, Research Director of the Division of Orthopaedic Surgery McGill University, Profesor of Surgery McGill University., Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CODIM-MBM-17-162
Record Dates: First submitted 2018-08-09; First posted 2018-09-24 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Total Knee Arthroplasty; Medial Pivot Knee Implant Design; Knee Joint Mechanics
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: A prospective, double-blinded, randomized control study consisting of a clinical follow-up followed by a knee kinematics assessment. Patients outcomes will be measured pre-operatively, and at 1 and 2 years post-surgery. Measures will include joint mechanics and neuromuscular activation during walking and stair stepping measured with motion capture and electromyography, and clinical/self assessment including pain in response to physical activity.
Who Masked: Participant, Outcomes Assessor
Masking Description: The Participants and the researchers at the Constance Lethbridge Rehabilitation Centre responsible for collecting the kinematic and gait data (motion capture, questionnaires, performance measures) will be blinded.
  For analysis purposes the Participants will be dummy coded (0 = one group, 1 = the other group). The blinded parties will know the dummy code but they will not know which group is assigned to each code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Zimmer MP Persona (Experimental): Zimmer MP Persona is total knee prosthesis intended to resurface the articulating surface of the femoral, tibial and patellar bones. It employs modular components between the tibial plates and articular surfaces and a medial congruent bearing manufactured from Vivacit-E Highly Crosslinked Polyethylene (HXPE). Persona® Medial Congruent Bearing is available in several sizes and offers up to a 13mm anterior lip height to provide greater anterior constraint and subluxation resistance. Can be used with a with both cruciate retaining and posterior stabilized femoral provisionals
  Interventions: Device: Zimmer MP Persona
- Zimmer Persona Knee-PS (Active Comparator): Zimmer Biomet Persona® Knee-PS is a semiconstrained knee prosthesis that employs modular components between the tibial plates and articular surfaces. The device is intended to resurface the articulating surface of the femoral, tibial and patellar bones. The posterior stabilized (PS) femoral provisionals and components can be used with the PS or constrained posterior stabilized (CPS) bearings provisionals and components when the PCL is deficient and removed.The Persona Femur offers 21 distinct profiles, in 2 mm increments.
  Interventions: Device: Zimmer Persona Knee-PS
- Healthy Participants (No Intervention): The control group for the kinematic assessment

INTERVENTIONS:
Device: Zimmer MP Persona — The medial pivot Persona® knee implant with a Medial Congruent™ Bearing
  Other Names: Medial Pivot Persona; Persona knee implant with a Medial Congruent Bearing
  Arms: Zimmer MP Persona
Device: Zimmer Persona Knee-PS — Persona the personalized knee system
  Arms: Zimmer Persona Knee-PS

SUMMARY:
Knee osteoarthritis (OA) is a highly prevalent condition that results in substantial pain and loss of function. The end stage treatment for knee OA is total knee arthroplasty (TKA), a common and safe procedure typically performed for relief of symptoms. However, an increasing number of patients are complaining about their TKA due to altered sensations between their previous joint and the implant. Although several designs have been proposed to improve these outcomes, the knee kinematics after TKA remains different from physiological kinematics. The Medial Pivot TKA design was introduced to closely mimic normal knee kinematics and create the natural feeling of the knee. This study is intended to evaluate the clinical effectiveness and ability to restore knee motion of two TKA devices: the Medial Pivot Persona TKA Zimmer design with the traditional Zimmer Persona Knee-PS. The investigator's hypothesis is that the Medial Pivot design will results in better patient outcomes and restore knee motion at natural parameters.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, randomized control study comparing the TKA Zimmer Medial Pivot Persona design to the traditional Zimmer Persona Knee-PS. Eighty patients requiring a TKA will be recruited and randomized to one of the two treatment arms following confirmation of eligibility criteria. Forty age and sex matched healthy participants with no knee OA will also be recruited to provide a comparator measure of "normal" joint motion.

Clinical follow-up visits and radiographic assessments will be performed pre- and post-operative at 6-weeks, 1-year, 2-years. Knee kinematics and self-assessment will be completed at the following intervals: pre-operative as baseline assessments for knee motion, 1-year, 2-years. Measures will include joint mechanics and neuromuscular activation during walking and stair stepping measured with motion capture and electromyography, and clinical/self assessment including pain in response to physical activity. Any other adverse events and complications (i.e, implant failure, re-operation, infection) will be record throughout the study.

Healthy participants will only be assessed once to provide normative data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with osteoarthritis, who in the opinion of the investigator, are suitable candidates for primary total knee replacement using the devices specified in the protocol;
* Males and females between 18 - 80 years at the time of surgery;
* Individuals who understand the conditions of the study and are willing and able to provide informed consent for participation in the study;
* Individuals who are willing and able to participate for the length of the prescribed term of follow-up;
* Individuals who are willing and able to complete all the assessments specified by the study protocol.

Exclusion Criteria:

* The presence of previous failed lower extremity arthroplasty or metalwork in situ;
* Patients with severe hip osteoarthritis;
* Patients with lower extremity trauma requiring surgery within 1 year;
* Patients with inflammatory arthritis, severe neurological conditions, or severe cardiovascular conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Knee mechanics | pre-operative (as baseline) and at 1 and 2 years following TKA
  nee motion will be assessed using 3-dimensional optical motion capture sampled at 100 Hz, floor and step mounted force plates sampled at 2000 Hz, and wireless 16-channel electromyography (EMG) system sampled at 2000 Hz.
  Knee motion trials will require participants to ambulate at self-selected speeds over 8 meters followed by complete step up/down trials on a 20 cm step. For step up, the surgical limb will be placed on the step to start while for step down, both limbs will start on the step. The order of step up and down trials will be randomized. Participants will perform 2 practice trials followed by testing. Testing will proceed until 5 successful trials of each activity are collected. They will be allowed 30 seconds of rest between trials.
  The primary motion capture variables will include principal component scores that capture changes in range of motion for knee rotation and flexion angles for each activity.

SECONDARY OUTCOMES:
Muscle activation | pre-operative (as baseline) and at 1 and 2 years following TKA
  Muscle activation will be measured by surface electrodes placed bilaterally over the following muscles: vastus lateralis and medialis, rectus femoris, lateral (biceps femoris) and medial (semitendinosus) hamstrings, and lateral and medial gastrocnemius. The isometric exercises will include: 1) knee extension in sitting with the knee in 45 degrees of flexion; 2) knee flexion in sitting with the knee at 55 degrees of flexion; 3) ankle plantarflexion in long sitting with the ankle in neutral; and 4) standing unilateral heel rise. Participants will perform 1 practice and 2 collection trials for each exercise. They will be allowed 30 seconds of rest between trials.
The 30 seconds Chair Test - Physical Function Performance Test | at 1 and 2 years following TKA
  Participants will be asked to complete "the 30 seconds Chair Test", a physical function performance test measuring the maximum number of sit-to-stand repetitions on a standard chair with a seat height = 46 cm.
The Stair Climb Test - Physical Function Performance Test | at 1 and 2 years following TKA
  After resting for 5 minutes, the participants will be asked to complete "the Stair Climb Test", a physical function performance test assessing the time [seconds] to ascend and descend a 11-step stair, each step 16 cm high.
The 6 Minutes Walk Test - Physical Function Performance Test | at 1 and 2 years following TKA
  After resting for 5 minutes, the participants will be asked to complete "the 6 Minutes Walk Test", a physical function performance test measuring the distance [meters] ambulate in 6 minutes. The participants will be allowed to rest during the test but the timer will not be stopped.
Knee Osteoarthritis and Outcome Score (KOOS) Self-Evaluation Questionnaire for Implant Performance | pre-operative (as baseline) and at 1 and 2 years following TKA
  Participants will be asked to complete the "Knee Osteoarthritis and Outcome Score (KOOS)" questionnaire. The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used, and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
EQ-5D-5L Self-Evaluation Questionnaire for Implant Performance | pre-operative (as baseline) and at 1 and 2 years following TKA
  Participants will be asked to complete the "EQ-5D-5L" questionnaire, a measure of health-related quality of life that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Global Rating of Change (GRC) Self-Evaluation Questionnaire for Implant Performance | pre-operative (as baseline) and at 1 and 2 years following TKA
  Participants will be asked to complete the GRC questionnaire to rate the improvement or deterioration over time compared to the pre-operative visit. The GRC is a 15-point scale (-7=Worse, +7=Better) to assess the participant current health status, recall that status at a previous time-point, and then calculate the difference between the two. The magnitude of this difference will be scored on a numerical or visual analogue scale.
Sensitivity to Physical Activity | at 1 and 2 years following TKA
  Sensitivity to Physical Activity will quantify the pain response to standardized physical activity. Participants will be required to rate their pain before and after each Physical Function Performance Tests using a 0 (no pain) to 100 (most pain imaginable) numeric rating scale. To determine the SPA for each test, the pain before the test will be subtracted from the pain after the test.
Radiographs | pre-operatively, intra operatively and at 6 weeks, 1 year and 2 years post-operatively
  Radiographs (anteroposterior hip to ankle, standing anteroposterior; standing lateral and patellar axial views) will be taken pre-operatively, intra operatively and at 6 weeks, 1 year and 2 years post-operatively as part of standard care. Radiographic evaluation will consist of the assessment of limb alignment, component position, and presence of radiolucencies or osteolysis. Longitudinal changes of posterior femoral condylar offset and the degree of posterior tibial slope after the surgery will be also determined.
Adverse Events | intra operatively and at 6 weeks, 1 year and 2 years post-operatively
  Adverse events and unplanned hospital visits will be tracked and documented. This includes wound related problems (infections), deep vein thrombosis, pulmonary embolism, stiffness, implant loosening, implant instability, re-operation or removal of any components for any reason.

OTHER OUTCOMES:
Maximum Voluntary Isometric Contractions (MVIC) | pre-operative (as baseline) and at 1 and 2 years following TKA
  Following gait trials, participants will complete a series of four maximum voluntary isometric contractions (MVIC) as follows: 1) knee extension in sitting with the knee in 45o of flexion; 2) knee flexion in sitting with the knee at 55o of flexion; 3) ankle plantarflexion in long sitting with the ankle in neutral; and 4) standing unilateral heel rise. MVIC exercises 1-3 will be performed on an isokinetic dynamometer. Participants will perform 1 practice and 2 collection trials for each exercise. They will be allowed 30 seconds of rest between trials. The MVIC will be used to normalize the amplitude of EMG waveforms.

CONTACTS AND LOCATIONS:
Overall Officials: John Antoniou, MD, PhD, Principal Investigator — Jewish General Hospital
Locations (3):
- Canada (3):
  - Montreal General Hospital, Montreal, PQ
  - Lethbridge-Layton-MacKay Rehabilitation Centre, Montreal, PQ
  - Jewish General Hospital, Montreal, PQ

IPD SHARING:
Plan to Share IPD: No